CLINICAL TRIAL: NCT02075554
Title: Efficacy and Safety of Expandable Spacer in the Treatment of Degenerative Disc Disease Using the Minimally Invasive Transforaminal Lumbar Interbody Fusion Surgical Approach
Brief Title: Study of an Expandable Interbody Device for the Lumbar Spine
Acronym: CALIBER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Globus Medical Inc (Industry)
Collaborators: Mt. Sinai Medical Center, Miami (Other); Carolina Neurosurgery & Spine Associates (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGC10-009-001-PL_H_2
Record Dates: First submitted 2014-02-04; First posted 2014-03-03 (Estimated); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Intervention Model Description: Lumbar interbody cages
Oversight: Data Monitoring Committee: No

ARMS (1):
- CALIBER (Other): 1 or 2 levels of DDD between L2 and S1, treated with transforaminal interbody fusion
  Interventions: Device: CALIBER

INTERVENTIONS:
Device: CALIBER — Expandable interbody spacer

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of CALIBER expandable spacer for the treatment of degenerative disc disease. Radiographic outcomes, intra-operative parameters, clinical outcomes, and patient satisfaction will be obtained from patients in this 2 year follow-up clinical study.

DETAILED DESCRIPTION:
Patients will be followed-up at 3weeks, 6 weeks, 3 months, 6 months, 12 and 24 months with X-rays and questionnaires to determine their satisfaction, healing, fusion and return to work status

ELIGIBILITY:
Inclusion Criteria:

* DDD at 1 or 2 levels between L2 and S1
* Between 18 and 80 years of age
* Unresponsiveness to documented non-surgical treatment modalities for a minimum of six months
* Ability to provide a signed Informed Consent

Exclusion Criteria:

* Trauma at level(s) to be fused
* Previous documentation of osteopenia, osteoporosis, or osteomalacia to a degree that spinal instrumentation would be contraindicated
* Immunosuppressive disorder
* History of substance abuse
* Any known allergy to a metal alloy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-07; Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Cohen, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - South Florida Spine Institute at Mt Sinai Medical Center, Miami Beach, Florida
  - Carolina NeuroSurgery and Spine Associates, Charlotte, North Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The protocol was approved to enroll 60 patients but only 58 patients were enrolled.
Groups:
- CALIBER: 1 or 2 levels of Degenerative Disc Disease between L2 and S1, treated with transforaminal interbody fusion
  CALIBER: Expandable interbody spacer
Period: Overall Study
Arm/Group | CALIBER
Started | 58
Completed | 43
Not Completed | 15
Not completed — Lost to Follow-up | 7
Not completed — Withdrawal by Subject | 5
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Population: Includes only those patients who completed the study
Arm/Group | CALIBER
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 12
Age, Continuous [Mean (Full Range); unit: years] | 54 [32 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Fusion and Disc Height Maintenance
Description: Inter-vertebral disc height in millimetres at 24 month follow up.
Time Frame: 24 months
Population: Not all patients had x ray images to measure at 24 month follow up. A total of 33 surgical levels were measured from 29 patients.
Measure: Mean (Full Range); unit: millimetres
Units Other Than Participants: Surgical Levels
Arm/Group | CALIBER
Number analyzed (Participants) | 29
Number analyzed (Surgical Levels) | 33
millimetres | 11.60 [8.62 to 15.60]

2. Primary Outcome: Fusion Assessment
Description: An assessment of the fusion status of surgically treated spinal levels.
Time Frame: 24 months
Population: Only 29 patients were available for fusion assessment at 24 months, for a total of 33 surgical levels.
Measure: Count of Units; unit: Surgical Levels
Units Other Than Participants: Surgical Levels
Arm/Group | CALIBER
Number analyzed (Participants) | 29
Number analyzed (Surgical Levels) | 33
Surgical Levels | 33

3. Secondary Outcome: Patient Self Assessment
Description: Oswestry Disability Index. A 10 item questionnaire with responses scored 0 to 5 and then presented as a percentage score from 0 to 100, with higher scores denoting more disability.
Time Frame: Upto 24 mo
Population: Not all patients completed the Oswestry Disability Index questionnaire at 24 month follow up, leaving 38 responses.
Measure: Mean (Full Range); unit: scores on a scale
Arm/Group | CALIBER
Number analyzed (Participants) | 38
scores on a scale | 18.79 [0 to 66]

4. Secondary Outcome: Visual Analog Scale for Back Pain
Description: A visual scale from 0 to 100 in which the patient responds with their pain level by marking on the line, higher as more severe pain.
Time Frame: 24 months
Population: 38 patients completed the question at 24 month follow up
Measure: Mean (Full Range); unit: score on a scale out of 100
Arm/Group | CALIBER
Number analyzed (Participants) | 38
score on a scale out of 100 | 10.71 [0 to 78]

ADVERSE EVENTS:
Time Frame: Subjects were assessed for adverse events by their physician over 24 months postoperative time period at each follow up point (Intraoperatively, 6 weeks, 3 months, 6 months, 12 months and 24 months postoperatively).
Arm/Group | CALIBER
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI may release for publication with Sponsor's prior approval.